CLINICAL TRIAL: NCT05446662
Title: The Effect of Complementary Care Model on Patient Outcomes in Patients With Coronary Artery Bypass
Brief Title: The Effect of Complementary Care Model on Patient Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ummuhan Yigid, principal investigator, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AIBU-KVC-UY-02
Record Dates: First submitted 2022-06-20; First posted 2022-07-07 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Nursing Caries; Music Therapy; Aromatherapy; Preoperative Care; Postoperative Care; Complementary Therapies
MeSH Terms: interventions — Music Therapy; Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): After randomization, the patients in the control group will be given pre- and post-operative nursing care without any intervention.
- case group (Experimental): Patients in the case group after randomization will choose one or more of the music therapy, aromatherapy, progressive relaxation exercises and massage therapies according to their health care needs.
  Interventions: Other: music therapy; Other: aromatherapy; Other: Progressive Relaxation Exercises; Other: Hand massage

INTERVENTIONS:
Other: music therapy — Patients participating in the study will be informed about the application of music therapy in the preoperative period. The patients who will take part in the music group are given 30 minutes the day before the surgery, and 30 minutes a day on the 1st and 2nd days after the surgery. Music that is selected by the researcher and grouped as relaxing music, classical music, sufi music and Turkish folk music will be played. The patients will be listened to the music with headphones that cover the whole ear, and the music will be adjusted to make them feel comfortable.
  Arms: case group
Other: aromatherapy — Patients participating in the study will be informed about the application of aromatherapy in the preoperative period. During this period, patients undergo elbow test (1 drop of lavender oil will be dripped onto the inside of the patient's elbow, after 20 minutes, it will be evaluated whether an allergic reaction has developed). Lavender oil as aromatic oil will be administered to the patients in the aromatherapy group in the form of inhalation. Lavender oil inhalation (1 drop of 0.1 cc) It will be applied by inhalation with gauze on which 3-4 drops of lavender oil are poured. 30 minutes before surgery. Aromatherapy will be applied four times with an interval of 30 seconds on the 1st and 2nd days before and after the surgery.
  Arms: case group
Other: Progressive Relaxation Exercises — Patients participating in the study will be informed about relaxation exercises in the preoperative period. Progressive relaxation training will be applied to the patients for 30 minutes once a day, on the day before the operation and on the 1st and 2nd days after the operation.
  Arms: case group
Other: Hand massage — Patients participating in the study will be informed about the application of massage therapy in the preoperative period. 10-15 minutes once in the preoperative period. And in the postoperative period, the 1st and 2nd days are 10-15 minutes. application will be carried out. Lavender oil (Lavandula Angustifolia) will be used in hand massage, sweet almond oil (Prunus Amygladus Sativa) will be used as essential oil.
  Arms: case group

SUMMARY:
The study will be carried out in Bolu Abant İzzet Baysal University İzzet Baysal Training and Research Hospital Cardiovascular Surgery Clinic between January 2022 and February 2023.

The population of the study will consist of patients who will undergo coronary artery bypass in a planned heart and meet the inclusion criteria.

The sample of the study will consist of patients who meet the inclusion criteria, volunteer to participate in the study, and whose written consent has been obtained.

To calculate the sample size of the study; NCSS Pass 11.0 program was used. According to the result calculated in this program, it was seen that a total of 60 people, 30 people in each group, should be reached for two groups and 99% power (α: 0.05).

With this study, it is aimed to increase the job satisfaction and quality of nurses as well as to increase the satisfaction of the patients in terms of nursing.

By presenting the Complementary Care Model to our country for the first time with this study; In this context, it was planned to determine the effects of music therapy, progressive muscle relaxation exercise, aromatherapy and massage on the outcomes (nausea, vomiting, sleep, anxiety, pain, complications and satisfaction) of coronary artery bypass graft patients.

DETAILED DESCRIPTION:
Patients in the post-randomization application group will choose one or more of music therapy, aromatherapy, progressive relaxation exercises and massage therapies according to the predisposing factors, facilitating factors and health care needs in choosing these applications according to the complementary care model.

Before the application, data will be collected from the patients with an introductory form containing the demographic data of the patients, Visual Pain Scale (VAS), and State Anxiety Scale.

Vital signs (systolic blood pressure, diastolic blood pressure, pulse, body temperature and respiratory rate) before and after the operation (10., 30. and 60. min), before and again on the 2nd and 3rd days after the operation. It will be measured and recorded after the application (10th, 30th, and 60th minutes).

After the preoperative practices, vital signs will be measured and the Surgery-Specific Anxiety Scale will be filled in by face-to-face interview method.

On the 1st and 2nd postoperative days, after each application, the VAS, the state anxiety scale, the visual comparison scale to evaluate the satisfaction level of the patients from the interventions after the 2nd postoperative day applications, and the Richard-Campell Sleep Scale to evaluate the night's sleep of the individual will be used.

Complications seen in the patient will be recorded on the patient follow-up form while the patients are discharged.

Routine pre- and post-operative nursing care will be given to the patients in the control group after randomization.

Data will be collected from the patients with an introductory form including their preoperative demographic data, Visual Pain Scale (VAS), and State Anxiety Scale.

Vital signs (systolic blood pressure, diastolic blood pressure, pulse, body temperature and respiratory rate) before and after the operation (10., 30. and 60. min), before and again on the 2nd and 3rd days after the operation. It will be measured and recorded after the application (10th, 30th, and 60th minutes).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone coronary bypass surgery with a beating heart-off pump,
* Those who are classified as I, II and III according to the system that the American Society of Anesthesiologists (ASA) classifies by evaluating patients according to their physical health status before surgery,
* Patients who do not have respiratory problems and are not allergic to plants
* Those without cognitive impairment,
* Those who can speak and communicate in Turkish and agree to participate in the study,
* Patients with a body mass ratio of 30 and below,
* Those who do not have chronic pain, alcohol, drug and substance addiction,
* Those who do not have Covid 19 disease,
* Patients with systolic blood pressure above 95 mmHg,
* It was planned to include patients who had planned surgery and did not develop complications during or after the surgery.

Exclusion Criteria:

* Patients undergoing coronary bypass surgery using a cardiopulmonary bypass machine,
* Those who are classified as ASA IV, V and IV,
* Patients who could not be reached before surgery,
* People with asthma and allergies to plants
* Those with mental disorders (psychosis, dementia, delirium),
* Hearing, vision, speech, smell disorders,
* Those who do not speak Turkish, cannot communicate and do not agree to participate in the research,
* Patients with a body mass ratio above 30,
* Those with chronic pain, alcohol, drug and substance addiction,
* Having had a covid 19 disease,
* Patients with systolic blood pressure below 95 mmHg,
* Patients who underwent emergency surgery and had serious complications during and after surgery will not be included in the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Anxiety | the day before surgery
  After the pre-operative nursing practices, the Surgical Anxiety Scale will be filled by face-to-face interview method. State Anxiety Scale; consists of 20 items. The highest score that can be obtained from the scale is 80, and the lowest score is 20. The higher the calculated total anxiety score, the higher the anxiety level of the person who completed the scale.
Distribution of systolic blood pressure of patients in case and control groups in intraoperative and postoperative period follow-ups | Change from Baseline Systolic Blood Pressure on intraoperative 10 minutes to 1 hours ; postoperative 10 minutes to 1 hours postoperative
  Measurement of systolic blood pressure of patients in the control and case groups in intraoperative and postoperative period follow-ups
sleep quality | 2nd day after surgery
  The Richard-Campbell Sleep Scale will be used to assess the patient's nighttime sleep.The scale is a 6-item scale that evaluates the depth of night sleep, the time to fall asleep, the frequency of awakening, the time to stay awake when awakened, the quality of sleep, and the noise level in the environment. Each item is evaluated with a visual analog scale technique and a chart between 0-100. Scores on the scale; A score of 0-25 indicates very bad sleep, and a score of 76-100 indicates very good sleep.
Change from pain on postoperative period | 10 minutes after music therapy/ aromatherapy/hand massage/progressive muscle relaxation exercises and Aftermusic therapy/ aromatherapy/hand massage/progressive muscle relaxation exercises 1st and 2nd day after surgery
  Visual analog Scale. It is a scale used to measure and monitor the severity of pain and is evaluated by the patient. The scale starts with the absence of pain (0) and ends with excruciating pain (10).
Distribution of diastolic blood pressure of patients in case and control groups in intraoperative and postoperative period follow-ups | Change from Baseline diastolic Blood Pressure on intraoperative 10 minutes to 1 hours ; postoperative 10 minutes to 1 hours postoperative
  Measurement of diastolic blood pressure of patients in the control and case groups in intraoperative and postoperative period follow-ups
Distribution of heart rate of patients in case and control groups in intraoperative and postoperative period follow-ups | Change from Baseline heart rate on intraoperative 10 minutes to 1 hours ; postoperative 10 minutes to 1 hours postoperative
  Measurement of heart rate of patients in the control and case groups in intraoperative and postoperative period follow-ups
Distribution of body temperature of patients in case and control groups in intraoperative and postoperative period follow-ups | Change from Baseline heart rate on intraoperative 10 minutes to 1 hours ; postoperative 10 minutes to 1 hours postoperative
  Measurement of body temperature of patients in the control and case groups in intraoperative and postoperative period follow-ups
Distribution of respiratory rate of patients in case and control groups in intraoperative and postoperative period follow-ups | Change from Baseline respiratory rate on intraoperative 10 minutes to 1 hours ; postoperative 10 minutes to 1 hours postoperative
  Measurement of respiratory rate of patients in the control and case groups in intraoperative and postoperative period follow-ups

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant Izzet Baysal Training and Research Hospital, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided